CLINICAL TRIAL: NCT00314223
Title: Identification of Gene Polymorphism in Patients With Sick Sinus Syndrome in Chinese Population in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Other Study IDs: DMR94-IRB-167
Record Dates: First submitted 2006-04-12; First posted 2006-04-13 (Estimated); Last update posted 2006-04-13 (Estimated); Status verified 2006-04

CONDITIONS: Sinus Arrhythmia
MeSH Terms: conditions — Arrhythmia, Sinus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Background: Sinus node dysfunction is a major cause of bradycardia necessitating pacemaker implantation. Evidences of genetic study supported that some genes involved in the pacemaker current or renin-angiotensin system were related to sinus node dysfunction. However, the influence of gene polymorphisms on sinus node dysfunction was not well studied.

Methods: A group of 100 patients with documented sinus node dysfunction and 100 age- and sex- matched healthy control patients will be enrolled into this study. Gene polymorphism study includes the angiotensin-I converting enzyme gene, angiotensin II type 1 receptor gene, HCN1-4, SCN5A, KCNE and other possible gene polymorphisms which are related to sinus node function based on previous reports. Genetic polymorphisms are identified with polymerase chain reaction-based restriction analysis. Comparison of multiple haplotype analysis and single-locus analysis will be analyzed between the cases and controls.

Estimated Results: Some genetic polymorphisms of these genes which are related to sinus node function or rennin-angiotensin system will show association with sinus node dysfunction. In multilocus haplotype analysis, some genetic haplotype profiles may demonstrate significant difference between cases and controls. In single locus analysis, some genetic polymorphisms may be associated with sinus node dysfunction.

Estimated Conclusion and Clinical Implication: This study will demonstrate the genetic polymorphisms in RAS genes or some other genes associated with sinus node dysfunction. These results will support the roles of these genetic polymorphisms in determining the risk of sinus node dysfunction among the Chinese population in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. Heart rate was less than 40/min or long pause more than 3 seconds in series EKG or 24-hour EKG.
2. Sinus nodal recovery time exceeds 1600 ms in cardiac electrophysiology study.

Exclusion Criteria:

1. Severe systemic disease.
2. Acute coronary syndrome.
3. Bradycardia with reversible cause.

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2006-02; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Yow Chen, MD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan